CLINICAL TRIAL: NCT06497907
Title: Prevalence of Environmental Enteropathy Among Infants and Children With Growth Faltering
Brief Title: Environmental Enteropathy Among Infants and Children With Growth Faltering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, Lecturer of pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 260/2021
Record Dates: First submitted 2024-06-25; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Growth Failure; Enteropathy
MeSH Terms: conditions — Failure to Thrive; Intestinal Diseases

STUDY DESIGN:
Intervention Model Description: Patient with growth faltering whose weight still below -2 SD for age and sex on the WHO scores after 12 weeks of nutritional rehabilitation with polymeric formula, underwent upper gastrointestinal endoscopy and who were diagnosed as environmental enteropathy, received nutritional rehabilitation with peptide based formula and probiotics
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with growth faltering (Experimental): Patient with growth faltering whose weight still below -2 SD for age and sex on the WHO scores after 12 weeks of nutritional rehabilitation with polymeric formula, underwent upper gastrointestinal endoscopy and who were diagnosed as environmental enteropathy, received nutritional rehabilitation with peptide based formula for 8 weeks and were reassessed.
  Interventions: Dietary Supplement: polymeric formula; Dietary Supplement: peptide based formula

INTERVENTIONS:
Dietary Supplement: polymeric formula — Patients with growth faltering received nutritional rehabilitation with polymeric formula and were reassessed after 12 weeks by anthropometric measurements
Dietary Supplement: peptide based formula — patients who were defined as non responders and underwent upper gastrointestinal endoscopy and diagnosed as environmental enteropathy, received nutritional rehabilitation with peptide based formula

SUMMARY:
The study was conducted on 200 patients with growth faltering on 2 phases. In the first phase the patient received nutritional rehabilitation with polymeric formula for 12 weeks then they were reassessed by anthropometric measurements and those whose weight remained below -2 SD for age and sex on the WHO scores were defined as non responders and entered the second phase. In the second phase Upper Gastrointestinal endoscopy was done and then patients received nutritional rehabilitation with peptide based formula and probiotics then were reassessed after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose weight below -2 SD for age and sex on the WHO scores.

Exclusion Criteria:

* Secondary cases of malnutrition or undernutrition.
* Patients with symptoms of GIT problems as chronic vomiting, chronic or bloody diarrhea, chronic abdominal distension, hematemesis or bleeding per rectum.
* Patients who can't commit to a follow up visit every two weeks.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Assessment of the prevalence of environmental enteropathy among children with faltering growth. | 12 weeks of nutritional rehabilitation with polymeric formula.
  Assess the number of patients whose weight still below -2SD and upper gastrointestinal endoscopy showed the criteria of environmental enteropathy.

SECONDARY OUTCOMES:
Determine the increase in weight of children with growth faltering and environmental enteropathy after nutritional rehabilitation with peptide-based formula. | 8 weeks of nutritional rehabilitation with peptide-based formula.
  Weight z- score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine-Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided